CLINICAL TRIAL: NCT03302000
Title: Early Visual Stimulation in Preterm Infants at Home From 0 to 3 Months
Brief Title: Visual Stimulation of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Adriana Neves Dos Santos, Professor, Reseacher, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UFSC-SIGPEX / 201610782
Record Dates: First submitted 2017-09-30; First posted 2017-10-04 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Preterm Infant
Keywords: prematurity; sensory stimulation; rehabilitation; infant
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2-arm, parallel-groups, pragmatic superiority randomised controlled trial. Allocation ratio will be 1:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two kind of researchers will be part of the study: a) assessors, which are the researchers that will perform assessments and apply stimulation with the caregivers; b) ratters, which are the researchers that will rate the scales from videos. Assessors will not be blind to group allocation. Ratters will be masked to group allocation, since videos analyses will be performed using coded study allocation. The statistician will also be blind to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual stimulation (Experimental): Early visual stimulation (EVS) will be implemented by caregivers.
  Three phases:
  1. the caregiver will establish eye-to-eye contact with the infant. The caregiver will communicate with the infant talking, singing, changing facial expressions, touching his/her face. Total duration of this part of stimulation is between 2 and 3 minutes
  2. the caregivers will present visual contrast cards at a distance of 15-20 centimetres
  3. the caregiver will present two toys to the infant
  Stimulation will last for 28 days (4 weeks) in total, one time a day for 10-15 minutes, all days week.
  Interventions: Other: Early Visual Stimulation; Other: standard care
- standard care (Other): Caregivers will receive an Illustrated Handbook, according to the age range of birth to three months. Assessors will explain all information contained in the handbook after the first assessment and randomisation.
  Interventions: Other: standard care

INTERVENTIONS:
Other: Early Visual Stimulation — Early visual stimulation
  Arms: Visual stimulation
Other: standard care — standard care

SUMMARY:
Introduction: Prematurity rate has increased and is a risk factor for developmental delay. Preterm infants with low visual tracking might present deficits in cognition, language, and fine motor function in future ages. Few studies applied home stimulation of the visual system for preterm infant (PT) at an early age.

Objective: To compare the effects of early visual stimulation to a standard care group in visual function, motor and sensory development.

Methods: Randomized controlled trial. At home setting. Thirty healthy preterm infants, gestational age from 28 to 37 weeks, aged from one to two months of corrected age at the entrance of the study, with low visual function, will be evaluated. Participants will be randomly allocated to: (1) a standard care group, receiving orientation about general sensory and motor development, (2) an early visual stimulation group receiving a 4-week home based protocol applied by caregivers additional to standard care. Outcomes will be measured at before the beginning of stimulation, at the end of stimulation and at 6 months of corrected age. Primary outcome is visual function evaluated by ML Leonhardt Battery of Optotypes. Secondary outcomes include motor and sensory development evaluated by scales.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 28 and 37 weeks
* age at enrolment between one to two months of corrected age t
* absence of visual impairments evaluated with Red Reflex Examination and complete ophthalmology exam, which will be performed by a doctor at the hospital or the basic health units where the infants will be recruited
* infants at home
* presence of low acuity assessed by the ML-Leonhardt Optotypes Battery (absence of alertness, fixation and attention in at least three cards, or visual tracking classified as absent or brief for more than three cards)

Exclusion Criteria:

* presence of any diagnosed neurological diseases
* presence of diagnosed respiratory diseases
* hypoxemia, hyperventilation or hypo-ventilation during assessments
* presence of congenital diseases
* presence of diagnosed visual impairments, such as blindness or low vision
* extreme premature, ie, with gestation age bellow 28 weeks due to higher risk of retinopathy of prematurity
* birth weight less than 1,000 grams due to higher risk of retinopathy of prematurity
* absence of alertness according with Precthl and Beintema
* preterm infant with unstable physiological conditions
* preterm infant receiving any kind of intervention such as physical therapy, occupational therapy, early intervention, aquatic stimulation, at the same time that our stimulation protocol is being applied since they can be confounders
* infants with medical fragility that prevent them to participate.

Ages: 1 Month to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Visual function - alertness, fixation, attention, tracking | change measure: first day - before intervention; after intervention at home (28 days)
  Visual acuity will be assessed with ML Leonhardt Battery of Optotypes (MLLBOS) scale. MLLBOS consists of 8 visual carts, with high-contrast visual images of 12X12cm. The scale evaluates alertness, attention, fixation and visual tracking. The evaluation will be recorded by a digital video camera. The camera will be positioned fixed to the infant's face.

SECONDARY OUTCOMES:
Sensory profile | change measure: first day - before intervention; after intervention at home (28 days); at 6 months of corrected age
  Infant Sensory Profile Scale (SPS) is a 125 item, norm-referenced, parent-report questionnaire. Sensory processing is divided in six items: general processing, auditory processing, visual processing, tactile processing, vestibular processing and oral sensory processing.
Motor Development | change measure: first day - before intervention; after intervention at home (28 days)
  Motor development will be assessed with Test of Infant Motor Performance (TIMP). It is a functional motor scale for newborn infants and infants under 4 months of age. Twenty-eight Observed Items examine spontaneously emitted movements, such individual finger, ankle and wrist movements. Thirty-one Elicited Items, scored on 5-, 6-, or 7-point ordinal scales, test infant's movement responses to placement in various spatial orientations and to interesting sights and sounds.
Motor Development | change measure: at 6 months of corrected age
  Motor development will be assessed with Alberta Infant Motor Scale (AIMS). The AIMS is a validated and reliable measure of infant's development. The assessors observe the spontaneous repertoire of infant's skills detected through 58 items grouped under four postures: prone (21 items), supine (9 items), sitting (12 items), and standing (16 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Catarina, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one year of study completion